CLINICAL TRIAL: NCT04427332
Title: Smell and Taste Disorders in COVID-19 Patients: Prospective Observational Study
Brief Title: Smell and Taste Disorders in COVID-19 Patients
Acronym: COVID-19 ORL
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19 ORL
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: covid19
Keywords: Coronavirus; sars-covid-2; coronavirus infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19 infection related patients: All subjects that had access to the "nasopharyngeal swabs" service of the hospital for the detection of the Sars-CoV-2 virus, both hospitalized and discharged from the hospital and not hospitalized, from mid-May to the end of June 2020, will be consecutively enrolled. It is assumed that 500 people will be recruited.
  Interventions: Other: Investigation of smell and taste disorders

INTERVENTIONS:
Other: Investigation of smell and taste disorders — The study consists of an epidemiological investigation by means of a prospective observational study with the aim of investigating the demographic and clinical factors related to the sense of smell and taste in patients with Sars Cov 2 infection.

SUMMARY:
This is a prospective monocentric observational study with the aim of investigating the demographic and clinical factors related to the smell and taste disorders in patients with Severe Acute Respiratory Syndrome - Coronavirus - 2 (Sars-Cov-2) infection.

DETAILED DESCRIPTION:
BACKGROUND:

Preliminary observational data collected by Otorhinolaryngologist at the San Gerardo Hospital in Monza and by literature evidenced that numerous patients suffering from Sars-CoV-2 infection had smell and taste disorders. The are many data in the literature but few validated studies are available. Furthermore, it is not yet known in these patients what factors are related to the presence of olfactory and gustatory symptoms.

The aim of the study is to identify the demographic and clinical factors related to the smell and taste disorders in patients with Sars-CoV-2 infection, to evaluate the evolution of symptoms with a follow-up and to evaluate which factors influence the improvement of that symptoms.

STUDY DESIGN:

The study will include patients diagnosed with Sars-CoV-2 infection who have been hospitalized in the COVID wards of the San Gerardo Hospital in Monza and non-hospitalized patients but that get access to the "nasopharyngeal swabs" service of the hospital for the detection of the Sars-CoV-2 virus.

The study includes 3 timepoints. After acquiring informed consent, patient will be contacted on the phone and he will be asked to answer a multiple or short-answer questionnaire (T0) aimed at collecting demographic and clinical data, in particular relating to the smell and taste disorders, which will take place approximately 24 hours after running the swab. Follow-up period will follow, which will require patients to be contacted and invited by the Investigator to repeat the telephone questionnaire respectively 1 month (T1) and 3 months (T2) from the first compilation (T0).

The following information will be collected and recorded on a paper CRF:

* registry collection (date of birth, gender at birth)
* origin of the subjects: hospitalized, not hospitalized
* pathological, pharmacological history, allergies, smoking, flu vaccination
* date of onset of COVID19 symptoms
* smell and taste symptoms and temporal correlation with systemic symptoms (fever, dyspnoea, headache, rhinitis, gastrointestinal symptoms, arthralgias, skin manifestations)
* date of regression of the smell and taste symptoms

STATISCAL ANALYSIS:

A logistic regression model is used to identify what the clinical and demographic factors associated with the onset of the disease of interest are.

The composite endpoint consisting of the presence of smell and / or taste disorders vs the absence of both pathologies will be used as a variable. The secondary analyzes will concern only the subjects who have declared that they have had the disease in the study and, through a logistic or ordinal regression model, we will try to identify which factors are associated with the positive evolution of the disease at T3 compared to T0.

ELIGIBILITY:
Inclusion Criteria:

1. The study should include patients diagnosed of Sars-Cov-2 infection carried out at the San Gerardo Hospital of Monza:

   * discharged from the COVID + wards of the San Gerardo Hospital in Monza
   * not hospitalized subjected to nasopharyngeal swab for Sars-Cov-2 at the San Gerardo Hospital in Monza:
2. Patients older than or equal to 18 years.
3. The informed consent that will be freely granted and acquired before the start of the study.

Exclusion Criteria:

1. Patients without ascertained diagnosis of Sars-Cov-2 infection carried out at San Gerardo Hospital in Monza;
2. Patients with previous or current documented rhinosinusal pathologies, previous rhinosinusal surgery, previous cranio-facial trauma, previous neurosurgical and maxillofacial surgery interventions conditioning neurological or sensorineural deficits at the rhinosinusal level, neuropsychiatric pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects belonging to the nasopharyngeal swabs service for the detection of the Sars-CoV-2 virus, both discharged from the hospital and not hospitalized, who will meet the inclusion / exclusion criteria, from mid-May until the end of June 2020 will be consecutively enrolled. It is assumed to recruit about 500 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Identification of demographic and clinical factors in covid19 patients. | Until patient discharge from the hospital (approximately four months)
  Identify the demographic and clinical factors related to the sense of smell and taste in patients with Sars-CoV-2 infection included in the study.

SECONDARY OUTCOMES:
Description of the disturbances of smell and taste | Until patient discharge from the hospital (approximately four months)
  Description in patients with Sars-CoV-2 infection the evolution of the symptoms (disturbances of smell and taste) understood as partial or total regression by 1-month and 3-month follow-up
Description of factors that influence smell and taste | Until patient discharge from the hospital (approximately four months).
  Define which factors (demographic and clinical) influence the improvement of the sense of smell and taste

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza-Ospedale San Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baig AM. Neurological manifestations in COVID-19 caused by SARS-CoV-2. CNS Neurosci Ther. 2020 May;26(5):499-501. doi: 10.1111/cns.13372. Epub 2020 Apr 7. No abstract available. PMID 32266761
- [Background] Hummel T, Whitcroft KL, Andrews P, Altundag A, Cinghi C, Costanzo RM, Damm M, Frasnelli J, Gudziol H, Gupta N, Haehne A, Holbrook E, Hong SC, Hornung D, Huttenbrink KB, Kamel R, Kobayashi M, Konstantinidis I, Landis BN, Leopold DA, Macchi A, Miwa T, Moesges R, Mullol J, Mueller CA, Ottaviano G, Passali GC, Philpott C, Pinto JM, Ramakrishnan VJ, Rombaux P, Roth Y, Schlosser RA, Shu B, Soler G, Stjarne P, Stuck BA, Vodicka J, Welge-Luessen A. Position paper on olfactory dysfunction. Rhinol Suppl. 2017 Mar;54(26):1-30. doi: 10.4193/Rhino16.248. PMID 29528615
- [Background] Fonteyn S, Huart C, Deggouj N, Collet S, Eloy P, Rombaux P. Non-sinonasal-related olfactory dysfunction: A cohort of 496 patients. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Apr;131(2):87-91. doi: 10.1016/j.anorl.2013.03.006. Epub 2014 Mar 26. PMID 24679542
- [Background] Klopfenstein T, Kadiane-Oussou NJ, Toko L, Royer PY, Lepiller Q, Gendrin V, Zayet S. Features of anosmia in COVID-19. Med Mal Infect. 2020 Aug;50(5):436-439. doi: 10.1016/j.medmal.2020.04.006. Epub 2020 Apr 17. PMID 32305563
- [Background] Nordin S, Bramerson A. Complaints of olfactory disorders: epidemiology, assessment and clinical implications. Curr Opin Allergy Clin Immunol. 2008 Feb;8(1):10-5. doi: 10.1097/ACI.0b013e3282f3f473. PMID 18188011
- [Background] Li YC, Bai WZ, Hashikawa T. The neuroinvasive potential of SARS-CoV2 may play a role in the respiratory failure of COVID-19 patients. J Med Virol. 2020 Jun;92(6):552-555. doi: 10.1002/jmv.25728. Epub 2020 Mar 11. PMID 32104915
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Derived] Galluzzi F, Rossi V, Bosetti C, Garavello W. Risk Factors for Olfactory and Gustatory Dysfunctions in Patients with SARS-CoV-2 Infection. Neuroepidemiology. 2021;55(2):154-161. doi: 10.1159/000514888. Epub 2021 Apr 1. PMID 33794531